CLINICAL TRIAL: NCT04820647
Title: A Strength-Based Intervention to Improve Job Interview Skills in Young Adults
Brief Title: KF STRIDE to Improve Job Interview Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Helen Genova, Associate Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1139-21
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kessler Foundation STRength IDentification and Expression (KF-STRIDE) (Experimental)
  Interventions: Behavioral: KF-STRIDE
- Services as Usual (No Intervention)

INTERVENTIONS:
Behavioral: KF-STRIDE — KF Stride works to improve identification (awareness) of personal character strengths and 2) express them in a socially appropriate way during a job interview
  Arms: Kessler Foundation STRength IDentification and Expression (KF-STRIDE)

SUMMARY:
The goals of the current study are to evaluate the preliminary effectiveness and feasibility of Kessler Foundation-Strength Identification and Expression (KF-STRIDE) in an 8-week randomized controlled trial comparing the intervention to services as usual (SAU).

DETAILED DESCRIPTION:
This study will evaluate the acceptability and effectiveness of a strength-based intervention (Kessler Foundation Strength Identification and Expression; KF-STRIDE) that can enhance job interview skills and employment. Despite possessing employable talents, the core social deficits of transition age youth with autism spectrum disorder (TAY-ASD) make it difficult for this group to articulate their individual strengths. This inability to identify and express one's strengths to a potential employer can negatively affect interview performance and lead to difficulty with job obtainment. Thus, the current proposal will examine the effectiveness (Aim 1), acceptability, usability, and feasibility (Aim 2) of a novel strength-based intervention, KF-STRIDE, which is designed to enhance the ability of TAY-ASD to identify personal strengths and effectively discuss them. The goals of the current study are to evaluate the preliminary effectiveness and feasibility of KF-STRIDE in an 8-week randomized controlled trial comparing the intervention to services as usual (SAU). The study will be performed at two private therapeutic schools. Compared to a SAU group, we hypothesize that the KF-STRIDE group will: a) improve the ability to identify strengths (Hypothesis 1), b) improve the ability to express strengths (Hypothesis 2), c) improve other job interview skills (Hypothesis 3) and finally c) improve ability to obtain employment 6-months following the intervention (Hypothesis 4). In this way, the current study is in line with the NIMH's experimental therapeutics model, as we will examine whether the intervention improves employment, as well as identify potential mechanistic targets that could affect outcome. In Aim 2, we will also monitor fidelity, acceptability, usability, and feasibility of the strength-based intervention. The long-term goal of the current research is to collect pilot data that will lead to fully-powered effectiveness and implementation evaluations of KF-STRIDE in other community settings.

ELIGIBILITY:
Inclusion Criteria:

* adolescents with Autism Spectrum Disorder
* Live in the United States of America
* Ages of 14-26
* Speak English fluently and at a 4th grade reading level

Exclusion Criteria:

* History of stroke, Traumatic Brain Injury, or neurological injury or disease in the past (like brain tumor or epilepsy).
* History of significant psychiatric illness
* Uncontrolled seizures or other unstable medical complications.

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Mock Job Interview | Week 8
  Blinded reviewers using a standardized scoring measure will rate the video recorded mock job interviews.
employment status (yes=1, no=0) | 6 months post intervention
  We will examine whether the person became employed or other changes to their employment status.
time-to-reach-employment (assessed as weeks since intervention completion). | 6 months post intervention
  We will examine how long it took for the person to obtain employment.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No